CLINICAL TRIAL: NCT05897736
Title: Analysis of Salivary Minerals Level Variations in Patients With Peri-implantitis
Brief Title: Salivary Minerals in Patients With Peri-implantitis
Acronym: mineral-perio
Status: Not yet recruiting | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Ivana Sutej, associate professor, University of Zagreb
Other Study IDs: 1-Mineral-Peri-Imp
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis; Peri-implant Mucositis; Periimplant Bone Loss; Periimplant Diseases; Peri-implant Health
Keywords: salivary minerals; peri-implantitis; peri-implant health; salivary biomarkers
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- peri-implant patient: Patients with diagnosed peri-implantitis

SUMMARY:
Patients included in the study will be recruited after arriving at the Faculty of Dentistry of the University of Zagreb. During the clinical examination, the patient's periodontal status (bleeding during probing, and the depth of the pockets around the implant) and a control x-ray will be taken to check bone loss. Saliva sampling will occur at 3-time points, when establishing the diagnosis of periimplantitis, before the start of therapy, and at the first control after treatment.

DETAILED DESCRIPTION:
Work protocol Through the Department of Oral Surgery and the Department of Periodontology, patients with symptoms of peri-implantitis are admitted for a planned intervention or radiological diagnostic-therapeutic procedure within the same day. The number of patients planned for inclusion in this research on changes in the level of salivary minerals in peri-implantitis is 25.

The treatment of peri-implantitis depends on the clinical symptoms, intra- and post-therapeutic complications are not expected, and a control examination is mandatory.

Patient screening Patient selection is based on social and medical criteria. Social criteria - the patient must understand the planned procedure and the postoperative course, agree to the procedure and giving a saliva sample.

Medical criteria - at the time of departure for the planned procedure, the patient's health must be in optimally stable condition if the patient suffers from chronic diseases.

The main clinical parameters are: 1. presence of plaque, 2. presence of BOP, 3. presence of pus, 4. increased probing depth, 5. loss of alveolar bone.

Preparation for the procedure On the day of the examination, the patient comes to the Institute at the agreed time, after which there is a short preparation and, in a pre-established order after a conversation with the researcher, a saliva sample is taken and a dental clinical examination is performed.

Before giving a saliva sample, patients should not eat, smoke or brush their teeth for at least 2 hours before.

Saliva sampling: Just giving a saliva sample is easy. The patient is placed in a quiet place, the method of spontaneous collection of unstimulated saliva is explained to him. Before the very beginning, he rinses his mouth with plain water, and a 5-minute stopwatch is started during which the patient spits the saliva that is produced in his mouth into a previously weighed polystyrene cup. After 5 minutes, the cup with saliva is placed in the freezer until further biochemical analysis, and the patient is referred for a clinical examination. Biochemical analysis: For the salivary minerals determination, a total of 200 μl of unstimulated saliva sample will be mixed with 40 μl of 5% lanthanum oxide and diluted with deionized water to 2.5 ml for atomic absorption spectrophotometry. Due to the strong affinity of calcium to form complexes with salivary proteins, non-centrifuged whole saliva containing both protein-bound and soluble calcium will be used for the assay. The measurements of salivary calcium will be performed by an atomic absorption spectrophotometer.

Clinical examination: the clinical examination will be performed with the help of a graduated periodontal probe. The clinical parameters that will be recorded are:

* Plaque index
* Bleeding after probing with a plastic probe (BOP)
* Supuration, secretion
* Probing depth greater than 3 mm
* Bone loss visible on X-ray.
* Clinical test of stability and mobility.
* The presence of swelling and redness of the mucous membrane
* foetor ex ore
* pain on percussion The treatment of periimplantitis depends on the state of the disease itself. Non-surgical therapy is indicated for peri-implant mucositis, while in the case of further progression of the disease and the appearance of pre-implantitis, non-surgical therapy is only an introduction to treatment, where surgical therapy is the main stage of treatment. For smaller bone defects, the method of choice for treatment is resective surgery, while for larger bone defects, regenerative surgical therapy is indicated.

A control examination is usually scheduled after six weeks. If the bleeding has stopped or decreased and if the probing depths (the depth of the "pockets" around the implant measured with a periodontal probe) have also decreased, the next control is scheduled as needed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed peri-implantitis

Exclusion Criteria:

* uncooperative patient
* younger then 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: •Patients who come for examination and treatment of the inflammatory process of a dental implant, peri-implantitis at School of dental medicine University in Zagreb. In order to confirm the diagnosis of peri-implantitis, the clinical criteria are as follows: • bleeding and/or suppuration during light probing; • probing depth of ≥ 3 mm; • loss of bone level ≥ 1 mm apical from the most coronary part of the intraosseous part of the implant.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in levels of salivary minerals with disease progression/regression | one year
  If it is shown that the minerals of bone metabolism change according to the direction of recovery, it is possible to use salivary minerals (calcium, magnesium and phosphates) as an aid in the prognosis of the course of recovery and reduce the time needed to make a decision on the type and intensity of therapy, as well as the loss itself and implant replacement